CLINICAL TRIAL: NCT06418737
Title: Sleep Hygiene Training in Gymnasts: Quasi-Experimental Study on Sleep Behaviour, Quality and Sleepiness
Brief Title: Sleep Hygiene Training in Gymnasts: Sleep Behaviour, Quality and Sleepiness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ümid Karlı, Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAIBU-SBF-UK-01
Record Dates: First submitted 2024-05-10; First posted 2024-05-17 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Sleep Hygiene; Habit, Good Sleep
Keywords: Sleep Quality; Sleep Hygiene; Sleep Habits; Athletes
MeSH Terms: conditions — Sleep Hygiene; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Single masked, randomized trial (experimental and control group)
Who Masked: Participant
Masking Description: Participants are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Training Group: (Experimental): Sleep Intervention: A 60-minute sleep hygiene education session will be delivered to the participants by an expert with experience in providing education in the areas of sports and sleep. Subsequently, interventions will be implemented to improve the sleep environments of the athletes who are staying at the facility
  Interventions: Behavioral: Sleep HygieneTraining
- Control Group (No Intervention): No training will be provided If offered by the control group participants, "sleep hygiene training" will be given after all the data collected from the Sleep Training Group

INTERVENTIONS:
Behavioral: Sleep HygieneTraining — Training Content
  * Importance of Sleep: The vital importance of sleep for physical and mental health.
  * Benefits of Adequate and Quality Sleep: The numerous benefits of sufficient and good quality sleep.
  * Sleep Stages: The different stages of sleep and their characteristics.
  * Sleep Hygiene: The concept of sleep hygiene and its importance for improving sleep quality.
  * What to Do?
  * What to Avoid for Better Sleep?
  Arms: Sleep Training Group:

SUMMARY:
Sleep is essential to human health and well-being. Lack of or poor sleep can negatively impact cognitive function, mood, and physical performance. Athletes, especially elite athletes, are at risk for sleep problems due to heavy training schedules and the stress of travel.

Lack of or poor sleep can negatively impact athletes in many ways, including lack of sleep can lead to mood disorders such as irritability, anxiety, and depression. This may have a negative impact on athlete motivation and participation in training. Sleep deprivation can lead to decreased muscle strength, endurance, and coordination. This can affect an athlete's performance in training and competition phase.

Sleep hygiene refers to a set of practices aimed at regulating the sleep environment and habits to improve sleep quality. Sleep hygiene education is an intervention designed to teach athletes about the importance of sleep hygiene to improve their sleep quality. As sleep quality improves, attention, concentration, memory, and decision-making skills also improve . This can help athletes to perform better during training and competition. As sleep quality improves, mood disorders such as irritability, anxiety, and depression decrease. This can increase athlete motivation and participation in training. As sleep quality improves, so does muscle strength, endurance, and coordination.

DETAILED DESCRIPTION:
This study will be one of the first study conduct on human to examine the effectiveness of sleep hygiene education among gymnasts. Gymnasts, like other athletes, are prone to sleep problems for the reasons mentioned above. Therefore, it is of great significance to study the impact of sleep hygiene education on the sleep quality of gymnasts and indirectly on sports performance and sleep health as well as its underlying mechanisms. Additionally, this study has the potential to make a significant contribution to the field of exercise science by examining the effectiveness of sleep hygiene education, specifically among gymnasts. By examining effects on sleep quality, athletic performance, and sleep health, this study could provide valuable insights into developing targeted interventions to optimize sleep and health in gymnasts.

The duration of the measurements will be in week 1 to see the acute effects of sleep, and as a minimum of 18-21 days is required for behavioural change, sleep measurements will be made in week 4.

ELIGIBILITY:
Inclusion Criteria:

* Voluntariness: Participants must be willing to participate in the study voluntarily and provide informed consent.
* Elite Gymnasts: Participants must be elite gymnasts competing at the national level.
* Being Healthy: Participants must be in good health and free of any significant medical conditions that could affect their sleep or participation in the study.
* No Prior Sleep Hygiene Training: Participants must not have received any formal sleep education or intervention in the past.

Exclusion Criteria:

* Complications During the Intervention: Participants who experience any complications during the sleep hygiene education intervention will be excluded from the study.
* Regular Use of Sleep-Affecting Medication

Ages: 15 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Male individuals will be included due to the fact that women's hormonal responses may cause heterogeneous findings and the difficulty in interpreting the findings due to their hormonal profile.
Enrollment: 14 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Actigraphy | Pre-test, following one week mid-test and following one month post-test
  Actigraphy is a less invasive method compared to other sleep measurement methods such as polysomnography
Athlete Sleep Behavior Questionnaire (ASBQ) | Pre-test and 1 month after the pre-test
  Athlete Sleep Behavior Questionnaire is a 17-item, Likert-type (1- Never, 5- Always) scale with 4 sub-factors (sports-related, sleep quality, habitual sleep efficiency, sleep disturbance)
Pittsburgh Sleep Quality Index (PSQI) | Pre-test and 1 month after the pre-test
  Pittsburgh Sleep Quality Index assesses various sleep-related factors, including sleep latency, sleep duration, sleep efficiency, and daytime sleepiness.
  It is a 19-item self-report questionnaire. Each item is scored from 0 to 3, and the total score ranges from 0 to 57. Higher scores indicate poorer sleep quality.
Cleveland Adolescent Sleepiness Questionnaire | Pre-test and 1 month after the pre-test
  Cleveland Adolescent Sleepiness Questionnaire provides a valid and reliable subjective measure of daytime sleepiness in adolescents.
  This Questionnaire consists of 16 items that measure daytime sleepiness. Scores range from 16 to 80 on a 5-point Likert scale (never: 1; rarely: 2; sometimes: 3; usually: 4; almost every day: 5). Five of the statements are scored in the reverse direction. Daytime sleepiness is obtained by summing the scores of the 16 items, and the higher the score, the higher the daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Umid Karli, PhD, Principal Investigator — Bolu Abant İzzet Baysal University, Faculty of Sport Sciences, Department of Coaching Education
Locations (1):
- Bolu Abant İzzet Baysal University, Faculty of Sport Sciences,, Bolu, Turkey (Türkiye)